CLINICAL TRIAL: NCT06507072
Title: Evaluating Adaptive Rock Climbing on Children With Upper Limb Differences
Brief Title: Adaptive Rock Climbing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Nina Lightdale, Principal Investigator, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-24-00150
Record Dates: First submitted 2024-07-05; First posted 2024-07-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Congenital Upper Limb Differences
Keywords: Adaptive sports; Rock climbing; Congenital Upper Limb Differences; Improved psychosocial health
MeSH Terms: conditions — Upper Extremity Deformities, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adaptive Rock Climbing (Experimental)
  Interventions: Behavioral: Adaptive Rock Climbing Program

INTERVENTIONS:
Behavioral: Adaptive Rock Climbing Program — Twelve week rock climbing program. The program will take place once per week over the course of twelve weeks.

SUMMARY:
The goal of this clinical trial is to assess changes in functional and psychosocial outcomes following a 12-week adaptive rock-climbing program for children with congenital upper limb differences. The main questions it aims to answer are

* Assess functional outcomes following a 12-week adaptive rock-climbing program.
* Assess psychosocial outcomes following a 12-week adaptive rock climbing program.
* Assess barriers to participation in adaptive sports.

Participants will complete 12-week adaptive rock climbing program.

ELIGIBILITY:
Inclusion Criteria:

* Parents 18 years and older.
* English or Spanish speaking.
* Participants with unilateral or bilateral congenital upper extremity disorders of limb formation differences ages 6-16.

Exclusion Criteria:

* Any patients younger than 6 years or older than 16 years, patients not fluent in English or Spanish, or patients with parents younger than 18 years.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Range of Motion at 12 Weeks | Baseline and 12 weeks
  An occupational therapist will measure the passive and active range of motion. These measurements will be conducted for the following: shoulder flexion, shoulder abduction, shoulder internal rotation, shoulder external rotation, elbow flexion/extension, forearm supination, forearm pronation, wrist extension, and wrist flexion. This will be measured in degrees.
Change from Baseline in KINDL Scores at 12 Weeks | Baseline and 12 weeks
  The KINDL questionnaire will be completed by both child and parent. It includes 24 Likert-scaled items associated with emotional well-being and self-esteem. Questionnaires will be scored according to instructions provided by KINDL.
Change from Baseline in Muscle Testing at 12 Weeks. | Baseline and 12 weeks
  Manual muscle testing will be measured by an occupational therapist. This will be measured from grade 0 to 5.
Change from Baseline in PROMIS Life Satisfaction Scores at 12 Weeks. | Baseline and 12 weeks
  To assess positive affect and well-being, children and parents will complete the PROMIS Pediatric Life Satisfactions v1.0 8-item Short Form. Patients will respond to statements such as "I was satisfied with my life," on a scale of 1 "Not at all" to 5 "Very much."
Change from Baseline in PROMIS Pediatric Global Health Scores at 12 Weeks | Baseline and 12 weeks
  To gain a general view of participants' perception of their own physical, emotional, and relational health, children will also be asked to complete the PROMIS Pediatric Global Health v1.0 7-item Short Form. Participants will respond to 7 statements on a scale of 5 "Excellent" to 1 "Poor."

SECONDARY OUTCOMES:
Assess Barriers to Participation in Adaptive Sports | At 12 weeks (post-intervention)
  Identify common transportation barriers through a demographic survey with transportation questions.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Lightdale, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No